CLINICAL TRIAL: NCT06892509
Title: The Effect of Mindfulness-Based Stress Reduction Programme (MBSR) on Quality of Life, Satisfaction With Life, Sleep Quality and Mental Well-Being of Menopausal Women: A Randomised Controlled Study
Brief Title: The Effect of Mindfulness Practice on Quality of Life, Life Satisfaction, Sleep Quality and Mental Well-being Levels in Menopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agri Ibrahim Cecen University (Other)
Collaborators: Ataturk University (Other)
Responsible Party: Principal Investigator, Ebru SOLMAZ, Lecturer, Agri Ibrahim Cecen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Atatürk Uni.
Record Dates: First submitted 2025-03-13; First posted 2025-03-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Mindfulness Based Stress Reduction
Keywords: Mindfulness-based stress reduction programme; Menopause; Mental well-being; Sleep quality; Life satisfaction; Quality of life
MeSH Terms: conditions — Psychological Well-Being; Sleep Initiation and Maintenance Disorders; Personal Satisfaction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Mindfulness-based stress reduction programme will be implemented
  Interventions: Behavioral: mindfulness-based stress reduction program
- No Intervention (No Intervention): Control group.The control group will not be treated for eight weeks.

INTERVENTIONS:
Behavioral: mindfulness-based stress reduction program — In this study, Mindfulness-Based Stress Reduction Programme will be applied to the women to be included in the experimental group as a nursing intervention. For this programme, the researchers participated in the Mindfulness-Based Stress Reduction Programme consisting of eight internationally validated modules consisting of eight sessions given by Tera Consultancy and completed the training. The certificates of the researchers are given in the appendices. The experimental group will receive a mindfulness-based stress reduction programme for a total of eight weeks, 2-1.5 hours per week. The mindfulness programme usually lasts eight weeks because it has been reported that this is an effective period of time to produce noticeable changes in brain structure, stress levels, emotional regulation and general well-being.
  Arms: Experimental

SUMMARY:
Although menopause is a normal physiological process in women's lives, it is often accompanied by physical and emotional symptoms that can negatively affect women's quality of life. Hot flushes and night sweats, physical discomfort, sleep disturbances, increased anxiety, irritability, depressive symptoms, fatigue are among the most common and disturbing menopausal symptoms. In order to have a healthy and happy menopause and postmenopausal period, reducing women's complaints during this period will improve their quality of life. Recently, women are increasingly turning to non-hormonal, complementary and alternative methods to improve their quality of life. One of these methods is mindfulness-based stress reduction programme. Studies examining the effects of mindfulness-based stress reduction programme on menopausal women are limited. Studies in Turkey have examined the effects of mindfulness-based stress reduction programme on quality of life, anxiety, depression and menopausal complaints, but there is no study on the effects on life satisfaction, sleep quality and mental well-being. This study aims to fill the gap in the literature by examining the effects of a mindfulness-based stress reduction programme on Turkish women. It was found that important parameters such as quality of life, life satisfaction, sleep quality and mental well-being decline during menopause. It is aimed to alleviate these problems with a mindfulness-based stress reduction programme and contribute to the active healthy aging process of women. The results of this study will contribute to the United Nations Sustainable Development Goals such as 'Healthy Individuals' and 'Gender Equality' by providing new strategies to improve the quality of life of menopausal women. It is also aimed to contribute to improving women's health and increasing the capacity of health services for active ageing by 2030. This study will be conducted on 90 women between the ages of 45-64 who have not had menstrual bleeding for at least one year and who volunteered to participate in the study, 45 of whom will be experimental and 45 of whom will be control, who applied to Ağrı Central Family Health Centre No. 6 in Ağrı province. The pre-test data of the women in the experimental and control groups, who were randomly assigned to the study, will be collected with the 'Descriptive Information Form', 'Utian Quality of Life Scale', 'Riverside Satisfaction with Life Scale', 'Pittsburgh Sleep Quality Scale' and 'Warwick-Edinburgh Mental Well-Being Scale'. The women in the experimental group will be given a mindfulness-based stress reduction programme. No intervention will be given to the control group. The post-test data will be collected from the women in the experimental and control groups after eight weeks. The data of the experimental and control groups (coded as X and Y) will be transferred to the computer environment by a statistician independent from the research and the data will be analysed and the findings will be reported.

DETAILED DESCRIPTION:
Experimental Group: Women in the experimental group will be given mindfulness-based stress reduction programme.

Control Group: No action will be taken.

Women who meet the inclusion criteria will be informed about the purpose, content and application of the study, and women in the experimental and control groups will be included in the study. At this stage, Personal Information Form, Utian Quality of Life Scale, Riverside Satisfaction with Life Scale, Pittsburgh Sleep Quality Scale, Warwick-Edinburgh Mental Well-Being Scale will be filled in both groups.

Informed consent will be obtained from the women at the end of the information process. Women will be assigned to the experimental and control groups using a simple randomisation table on the website www.random.org. Personal Information Form, Utian Quality of Life Scale, Riverside Satisfaction with Life Scale, Pittsburgh Sleep Quality Scale, Warwick-Edinburgh Mental Well-Being Scale will be applied to both groups. Women in the experimental group will also be given mindfulness training.

ELIGIBILITY:
Inclusion Criteria:

* Who agreed to participate in the research,
* Can read and write Turkish,
* Not diagnosed with a psychiatric illness,
* 45-64 years of age with no menstrual bleeding for at least one year,
* Using any CAM method (such as Reiki, phytoestrogens, acupressure),
* Women who score above 5 points on the Pittsburgh Sleep Quality Scale will be included.

Exclusion Criteria:

* Voluntary withdrawal from the research,
* Taking antidepressants, antihistamines, benzodiazepines, hypnotics, narcotics, etc,
* Women who started to use any CAM method (such as Reiki, phytoestrogens, acupressure) will be excluded from the study.

Ages: 45 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women in menopause
Enrollment: 86 (Actual)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Utian Quality of Life Scale | This form will be collected on day 1. The experimental group will be given mindfulness-based stress reduction training for 2 months. After the trainings are completed, the form will be applied again.
  It consists of four sub-dimensions. These are emotional quality of life sub-dimension, sexual quality of life sub-dimension, occupational/work quality of life sub-dimension and health quality of life sub-dimension. Each item of the scale is in five-point Likert type and the statements are ranked from 1 to 5 according to their suitability for the person. In the scale statements, 'strongly disagree' is evaluated on a scale of 1, 'disagree' on a scale of 2, 'somewhat agree' on a scale of 3, 'agree' on a scale of 4, and 'strongly agree' on a scale of 5. The scale consists of straight and reverse question items. The 4th, 7th, 7th, 8th, 11th, 12th, 12th, 13th, 15th and 16th question items of the scale are straight, a
Riverside Satisfaction with Life Scale | This form will be collected on day 1. The experimental group will be given mindfulness-based stress reduction training for 2 months. After the trainings are completed, the form will be applied again.
  In the scale consisting of a total of 6 questions, each question is scored from 1 to 7. The scale is a seven-point Likert type. In the scale statements, the expression 'strongly disagree' is evaluated over 1 point, 'moderately disagree' is evaluated over 2 points, 'slightly disagree' is evaluated over 3 points, 'neither agree nor disagree' is evaluated over 4 points, 'slightly agree' is evaluated over 5 points, 'moderately agree' is evaluated over 6 points, and 'strongly agree' is evaluated over 7 points. The scale is one dimensional. All items of the scale are positive, there is no reverse statement. Total scores ranged from 6 to 42, with higher scores indicating higher levels of life satisfaction.
Pittsburgh Sleep Quality Scale | This form will be collected on day 1. The experimental group will be given mindfulness-based stress reduction training for 2 months. After the trainings are completed, the form will be applied again.
  The index consists of 24 questions in total and each question is scored from 0 to 3. In the index, there are five questions asked for clinical information that are not used in the scoring to be answered by the bed mate of the individuals. In the index consisting of seven components; subjective sleep quality, habitual sleep efficiency, time to fall asleep, sleep duration, sleep disturbance, sleep medication use and daytime dysfunction are evaluated. The sum of the scores obtained from the seven components gives the total score of PDQI and the total PDQI score can be a score between 0-21. The sleep quality of individuals with a PDQI total score of 5 points or less is considered as 'good',
Warwick - Edinburgh Mental Well-being Scale | This form will be collected on day 1. The experimental group will be given mindfulness-based stress reduction training for 2 months. After the trainings are completed, the form will be applied again.
  This scale is a tool used to assess the mental well-being levels of individuals. The scale consists of 14 items and is 5-point Likert type. In the scale statements, 'never' is expressed as 1, 'rarely' as 2, 'sometimes' as 3, 'often' as 4 and 'always' as 5 points. Scale scores vary between 14 and 70 and there are no reverse items in the scale. There are no sub-dimensions in the scale. It is also stated that the increase in the scale scores is related to the increase in the mental well-being of the individuals.

CONTACTS AND LOCATIONS:
Locations (1):
- AgriIbrahimCecenU, Ağrı, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No